CLINICAL TRIAL: NCT06901947
Title: The Effect of Preoperative Oral Carbohydrate Solution Administration of Insulin Resistance in Patients Undergoing Elective Open-Heart Surgery
Brief Title: Carbohydrate Loading on Insulin Resistance in Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Jefferson K Hidayat, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes060
Record Dates: First submitted 2024-07-15; First posted 2025-03-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Investigator
Masking Description: Investigator is blinding to the intervention given to the subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mineral water (No Intervention): Patient is given mineral water 2 hours before operation
- Glucose Drink (Experimental): Patient is given glucose water 2 hours before operation
  Interventions: Dietary Supplement: Glucose drink

INTERVENTIONS:
Dietary Supplement: Glucose drink — Intervention group will receive maltodextrin glucose drinks 2 hours prior to the operation
  Arms: Glucose Drink

SUMMARY:
This study is a single-blind randomized clinical trial involving 40 adult patients undergoing elective open-heart surgery. The sample was allocated into two groups: 20 subjects in the oral carbohydrate fluid group and 20 subjects in the water group consumed 2 hours before surgery. Insulin resistance was measured by blood glucose levels, HOMA-IR index, and insulin tolerance tests. Postoperative outcomes were assessed by ICU stay duration, ventilator use, and hospital stay duration. Patient comfort factors were measured by hunger, thirst, nausea, and comfort levels.

DETAILED DESCRIPTION:
In general, preoperative fasting is mandatory for any kind of operations. This is intended to reduce the risk of aspiration during anesthesia procedure. According to recommendation from American Society of Anesthesiologist (ASA), fasting time limit is 8 hours for high calories food, 6 hours for moderate calories food, 4 hours for breastmilk, and 2 hours for clear fluid. Until today, many studies have shown that conventional fasting causes metabolic burden. Lengthy fasting period induces body's stress response, seen in increase in catabolic reaction, elevated contra insulin hormones such as glucocorticoid and catecholamine. In addition to that, surgical stimulus heightens this metabolic reaction which leads to insulin resistance. Insulin resistance causes hyperglycemia, which have a negative impact postoperatively. Several postoperative outcomes have been linked to insulin resistance, such as longer duration of ventilator and hospital stay, as well as the likelihood of postoperative infection. Cardio thorax surgery, as many other major surgeries pose a significant risk of metabolic derangement. Hyperglycemia is known to cause oxidative stress. As the risk of postoperative increases, the mortality and morbidity also increase. In the era of enhanced recovery after surgery, carbohydrate loading is given 2 hours before operation in attempt to improve outcome. Giving 50-250 grams of carbohydrate is expected to suppress catabolic process that usually occurs due to prolonged fasting. This strategy has been implemented in non cardiac surgery, which has shown benefit postoperatively. However, until today there are still limited studies regarding the use of carbohydrate loading on open heart surgeries. The investigators intend to evaluate the benefit of this practice on insulin resistance.

This study was a single-blind randomized clinical trial. The study took place in heart center of Ciptomangunkusumo (RSCM) Hospital and Jakarta Hear Center (JHC) Hospital, for 10 months starting from January 2023 to October 2023. Forty subjects were recruited following the approved ethical clearance by Ethics Committee, Universitas Indonesia. The investigators had a consecutive sampling with inclusion criteria of adult patients aged 18-65 years old who undergo open heart elective surgery and give their consent. The exclusion criteria are those with diabetes mellitus, gastroesophageal reflux, digestive malignancy, dementia, mental disturbances, as well as ASA classification of 4 or more. The drop out criteria applied were those who passed away during operation, experienced hypoglycemia with blood glucose < 70 mg/dl, withdrew from the research, and were not able to finish the data sampling.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18-65 years old undergoing elective open heart surgery
* Subjects giving informed consent

Exclusion Criteria:

* Subjects with diabetes mellitus
* Subjects with gastroesophageal reflux
* Subjects with digestive malignancy
* Subjects with dementia
* Subjects with mental health
* Subjects with ASA 4 or more

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Insulin resistance difference between two groups | Within 30 minutes before and 30 minutes after operation
  Insulin resistance seen in the level of blood glucose (mg/dL)
Insulin resistance difference between two groups | Within 30 minutes before and 30 minutes after operation
  Insulin resistance seen in the level HOMA-IR (unitless)
Insulin resistance difference between two groups | Within 30 minutes before and 30 minutes after operation
  Insulin resistance seen in the level insulin sensitivity test (%/minute)
Operation outcome difference between two groups | From completion of operation to ICU discharge or death, usually under 28 days
  Operation outcome in form of length of stay in the ICU (days)
Operation outcome difference between two groups | From completion of operation to hospital discharge or death, usually under 28 days
  Operation outcome in form of length of stay in the hospital (days)
Operation outcome difference between two groups | From completion of operation to cessation of ventilator use or death, usually under 28 days
  Operation outcome consists of duration of ventilator use (days)
Subjective well being difference between two groups | Preoperatively in the preparation room, usually around 1 hour before operation
  Subjective well being in form of hunger (Yes or No)
Subjective well being difference between two groups | Preoperatively in the preparation room, usually around 1 hour before operation
  Subjective well being in form of thrist (Yes or No)
Subjective well being difference between two groups | Preoperatively in the preparation room, usually around 1 hour before operation
  Subjective well being in form of nausea (Yes or No)
Subjective well being difference between two groups | Preoperatively in the preparation room, usually around 1 hour before operation
  Subjective well being in form of comfort (Yes or No)

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No